CLINICAL TRIAL: NCT02460237
Title: Pilot Testing an HPV Self-Test Intervention: A Novel Strategy for Reducing Cervical Cancer in Appalachia
Brief Title: HPV Self-Test Intervention in Ohio Appalachia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Paul Reiter, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: OSU-14282; NCI-2015-00726 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2015-05-28; First posted 2015-06-02 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Cervical Carcinoma; Human Papillomavirus Infection
Keywords: HPV
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections | interventions — Mass Screening; Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (intervention) (Experimental): Participants receive a study kit that includes culturally appropriate instructions for using and returning the HPV self-test device and a photo story information sheet about HPV and HPV self-testing. Participants are asked to complete the HPV self-test and return the test for HPV testing.
  Interventions: Procedure: Disease Screening; Other: Educational Intervention; Other: Laboratory Biomarker Analysis; Other: Survey Administration
- Arm II (control) (Active Comparator): Participants receive a study kit that includes standard instructions for using and returning the HPV self-test device and a standard information sheet about HPV and cervical cancer. Participants are asked to complete the HPV self-test and return the test for HPV testing.
  Interventions: Procedure: Disease Screening; Other: Informational Intervention; Other: Laboratory Biomarker Analysis; Other: Survey Administration

INTERVENTIONS:
Procedure: Disease Screening — Complete HPV self-test
  Other Names: Disease Screening Procedure; Screening; Screening Intervention
Other: Educational Intervention — Receive culturally appropriate instructions for using and returning the HPV self-test device and a photo story information sheet about HPV and HPV self-testing
  Other Names: Education for Intervention; Intervention, Educational
  Arms: Arm I (intervention)
Other: Informational Intervention — Receive standard instructions and information sheet
  Arms: Arm II (control)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Survey Administration — Ancillary studies

SUMMARY:
This study will pilot test a culturally appropriate human papillomavirus (HPV) self-test intervention among women from Ohio Appalachia in order to determine the feasibility of HPV self-testing as a potential cervical cancer screening strategy. The intervention group will receive culturally appropriate materials and the control group will receive standard materials with their HPV self-test device.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of HPV self-testing as a potential cervical cancer screening strategy and obtain preliminary efficacy data of culturally appropriate materials on self-test use.

OUTLINE:

Participants are randomized to 1 of 2 arms.

ARM I: Participants receive a study kit that includes culturally appropriate instructions for using and returning the HPV self-test device and a photo story information sheet about HPV and HPV self-testing. Participants are asked to complete the HPV self-test and return the test for HPV testing.

ARM II: Participants receive a study kit that includes standard instructions for using and returning the HPV self-test device and a standard information sheet about HPV and cervical cancer. Participants are asked to complete the HPV self-test and return the test for HPV testing.

Participants are followed up at 4 weeks for return of their HPV self-test device and then for 2 months after notification letters are sent.

ELIGIBILITY:
Inclusion Criteria:

* Ages 30-65
* No Pap test in the last 3 years
* Resident of an Ohio Appalachia county
* Not currently pregnant or was not pregnant in the last 3 months
* No history of invasive cervical cancer
* No history of hysterectomy; women will not be eligible for the pilot randomized controlled trial (RCT) if they participated in the focus groups that helped develop this study (focus groups were institutional review board [IRB] approved as Protocol 2014C0086) or the preliminary device test; we will also require women to read and understand English and have the ability to provide informed consent, which will be inferred upon completion and return of the study eligibility, consent, and Health Insurance Portability and Accountability Act (HIPAA) forms

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-06-14 (Actual); Study Completion 2017-03-15 (Actual)

PRIMARY OUTCOMES:
The proportion of women who return HPV-self tests | Up to 4 weeks from kit distribution
  A chi-square test will be used to test for a difference between the two groups.

SECONDARY OUTCOMES:
Attendance at a follow-up health care visit after HPV testing notification letters are sent (attended or did not attend) | Up to 2 months after notification letters are sent
  Descriptive statistics (e.g., proportions) will be calculated for the entire sample and by study arm.
Prevalence of HPV infection | After shipping the specimen, an expected average of 6 weeks
  Descriptive statistics (e.g., proportions) will be calculated for the entire sample and by study arm.
Specimen adequacy (whether participants self-collected an adequate specimen [yes or no] to allow for HPV testing) | After shipping the specimen, an expected average of 6 weeks
  Descriptive statistics (e.g., proportions) will be calculated for the entire sample and by study arm.

OTHER OUTCOMES:
Receipt of a Pap test (received or not received) | Up to 2 months after receiving notification letters are sent
  Descriptive statistics (e.g., proportions) will be calculated for the entire sample and by study arm.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Reiter, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Reiter PL, Shoben AB, McDonough D, Ruffin MT, Steinau M, Unger ER, Paskett ED, Katz ML. Results of a Pilot Study of a Mail-Based Human Papillomavirus Self-Testing Program for Underscreened Women From Appalachian Ohio. Sex Transm Dis. 2019 Mar;46(3):185-190. doi: 10.1097/OLQ.0000000000000944. PMID 30461597
- See also: The Jamesline — http://cancer.osu.edu